CLINICAL TRIAL: NCT04596891
Title: Feasibility Pilot of Acceptance and Mindfulness Based Exposure Therapy for Survivors of Cardiac Arrest
Brief Title: Acceptance and Mindfulness Based Exposure Therapy for Survivors of Cardiac Arrest
Acronym: AMBET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Yuval Y Neria, Professor of Medical Psychology, Research Foundation for Mental Hygiene, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8017
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: PTSD; Cardiac Arrest
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Heart Arrest | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Remotely delivered psychotherapy combining exposure therapy with mindfulness
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Eight sessions of exposure therapy combined with mindfulness delivered via videoconferencing platform.

SUMMARY:
The primary goal of this uncontrolled pilot trial is to examine feasibility, acceptability, safety, and preliminary efficacy of a new behavioral treatment for survivors of sudden cardiac arrest with clinically elevated symptoms of post-traumatic stress disorder (PTSD). Participants will be recruited among cardiac arrest survivors enrolled in the observational CANOE research study (CUIMC IRB# AAAR8497). Study participants will be interviewed about their symptoms and evaluated for baseline assessment before receiving eight weekly sessions of an acceptance and mindfulness-based exposure therapy (AMBET). Participants will be additionally evaluated at treatment mid-point (week 4), and at the end of treatment.

The treatment and all assessments will be conducted remotely via Zoom. To assess whether patients' physical activity is improved over the course of treatment, participants will be provided with a wearable device (Fitbit wristband) to monitor their physical activity.

The specific aims of this study are to: (1) develop an acceptable protocol for an AMBET intervention for survivors of sudden cardiac arrest with elevated PTSD symptoms (2) examine its safety and feasibility in a small sample of 14 patients (3) investigate acceptability and feasibility of the assessments and measurements including physical activity.

DETAILED DESCRIPTION:
Clinically elevated levels of PTSD symptoms occur in approximately 1 in 3 cardiac arrest survivors with intact cognitive function and are associated with increased risk for future cardiac events and mortality. Survivors of acute cardiovascular events are typically encouraged to monitor for somatic cues of cardiovascular activity that might indicate recurrent events. However, threat-related attention bias is a common sequela of trauma. In cardiac patients, this hypervigilant attention to interoceptive cues of danger may serve to maintain threat perception, as arousal amplifies awareness of internal stimuli. Elevated PTSD symptoms have also been associated with low adherence to physical activity and medication regiments in patients with elevated PTSD symptoms after other types of cardiovascular events in part because they can serve as traumatic reminders. Although several well-studied, validated treatments for PTSD exist, there is no evidence-based treatment for PTSD in cardiac arrest survivors. Standard PTSD interventions targeting fear extinction and threat perception in the context of current safety pose a problem in a population that is living with an actual ongoing cardiac threat. Thus, the investigators will be developing a de novo protocol for an Acceptance and Mindfulness-Based Exposure Therapy (AMBET) intervention that targets increased discriminatory perception through mindful interoceptive attention and adaptive threat responding. Initial evidence has been published to suggest the safety and potential efficacy of imaginal exposure in cardiac patients to reduce PTSD symptoms. Among PTSD treatments, exposure therapy is the most widely recommended. However, the efficacy is moderate, and high dropout rates are well documented. An innovative line of PTSD therapies can be found among mindfulness- and acceptance-based treatments. Although large scale RCTs are still limited, there are promising findings of treatment effects on reduced PTSD symptoms. Reported dropout rates have been low across treatments, indicating a high degree of treatment acceptability. The addition of mindfulness components to exposure therapy has been proposed to enhance the effects of exposure as well as the willingness to engage in them. Of particular interest for cardiac patients are findings that mindfulness-based approaches have normalized cortisol levels and reduced inflammatory biomarkers in PTSD patients, as these are physiological processes that have been implicated in the links between PTSD and cardiovascular risk. Several mechanisms have been posited to underlie the efficacy of mindfulness-based approaches including increased metacognitive awareness of interoceptive sensations and mind-body connections. Furthermore, and contrary to the associations found between hypervigilant interoceptive awareness and psychopathology, mindful attention to interoceptive cues has been linked with adaptive, resilience-enhancing behaviors. The goals of the AMBET treatment will be to reduce PSTD symptoms and hypervigilance to internal stimuli (i.e., interoceptive bias), and increase cardiovascular health behaviors (medication adherence, physical activity) following cardiac arrest. Following psychoeducation about PTSD and cardiovascular disease related health behaviors, participants will be engaged in in-vivo and imaginal exposure exercises to reduce avoidance responses. Participants will be introduced to acceptance and mindfulness-based strategies that will be practiced in session and as homework assignments. Eight 90 minute sessions will be delivered to patients individually on a weekly basis through HIPAA-compliant zoom-hosted video visits. Patient symptoms will be assessed by an independent evaluator before, at mid-point, and post-treatment. A within-subjects repeated measures design will be used to assess the feasibility of conducting all aspects of the study remotely, including recruitment, assessment, and treatment delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the age of 18-85
2. A PCL-5 score of ≥ 33 at most recent assessment (≥ 30 days post cardiac arrest)
3. Hospitalization for cardiac arrest with cardiac etiology at any time in the past.

Exclusion Criteria:

1. Heart failure with severe systolic dysfunction (ejection fraction ≤ 25%)
2. Terminal non-cardiovascular illness with life expectancy <1 year
3. History of psychiatric diagnosis of psychotic episode, psychotic disorder, schizophrenia, schizoaffective disorder
4. Current severe depression determined by a) a score of >25 on the Hamilton Rating Scale for Depression (HAM-D-17-item), and b) clinical assessment.
5. Significant cognitive impairment defined by Cerebral Performance Category Score ≥3, and/or MMSE score of <24 neurological impairment precluding ability to complete study questionnaires.
6. Active suicidal ideation or behavior.
7. Current primary diagnosis of bipolar disorder.
8. Current unstable or untreated medical illness.
9. Current drug or alcohol misuse: severe alcohol/cannabis or any other substance use disorder (except nicotine).
10. Recent psychotropic medication change or initiation within the last 3 months.
11. Initiation of other psychotherapy within the last 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Neria, PhD, Principal Investigator — Columbia University and NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Bergman M, Markowitz JC, Kronish IM, Agarwal S, Fisch CT, Eder-Moreau E, Neria Y. Acceptance and Mindfulness-Based Exposure Therapy for PTSD After Cardiac Arrest: An Open Feasibility Trial. J Clin Psychiatry. 2023 Nov 22;85(1):23m14883. doi: 10.4088/JCP.23m14883. PMID 38019593

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.55 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Diagnosis at Baseline: Posttraumatic Stress Disorder (PTSD) [Count of Participants; unit: Participants] | 11
Diagnosis at Baseline: Depression [Count of Participants; unit: Participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Symptoms Over Time
Description: Reduction in symptoms as measured by the Clinician Administered PTSD Scale (Caps-5: ranging from 0-80 ) from pre- to post-treatment. Lower scores mean better outcome (reduction of symptom severity).
Time Frame: Baseline, At 4 weeks, Post-treatment: approximately 3 months from intake
Population: Baseline, midpoint, and post-treatment analysis of symptom scores for participants who completed the study protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
score on a scale
  Baseline | 37.00 (7.05)
  Midpoint (4 weeks) | 25.90 (9.15)
  Posttreatment | 16.20 (10.84)
Statistical Analysis 1: Comparison: Intervention; No control group, open trial for feasibility/safety; Test type: Other — Repeated measures ANOVA; p < 0.001, ANOVA; F ratio = 20.62 — The F ratio is used to evaluate the main effect of time in the ANOVA in relation to the critical F ratio
Statistical Analysis 2: Comparison: Intervention; Test type: Other — Paired-samples t-test (baseline to post-treatment); p = 0.002, t-test, 2 sided; paired-samples t-test = 5.2, 95% CI 2-sided [-1.79 to 12.93]

2. Primary Outcome: Change in Medication Adherence Over Time
Description: Participants' cardiac medication adherence is measured by self-report using the Morisky Medication Adherence Scale (MMAS). Scores can range from 0-8. If a patient scores higher on the scale, they are evaluated as more adherent.
Time Frame: End of treatment: approximately 3 months from intake
Population: baseline conducted on all enrolled participants, posttreatment data available for 9 patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 11
score on a scale
  Baseline | 3.18 (1.83)
  Posttreatment: number analyzed (Participants) | 9
  Posttreatment | 2.38 (1.41)

3. Primary Outcome: Change in Physical Activity Over Time
Description: Participants level of physical activity is measured objectively by a wrist worn Fitbit device.
Time Frame: End of treatment: approximately 3 months from intake
Measure: Mean (Standard Deviation); unit: daily steps
Arm/Group | Intervention
Number analyzed (Participants) | 11
daily steps
  Baseline | 7109.83 (5377.75)
  Posttreatment | 9296.83 (5600.44)

4. Secondary Outcome: Participant Satisfaction With Treatment
Description: Treatment satisfaction will be measured by the Client Satisfaction Questionnaire (CSQ-3). Scores range from 0-12 with higher scores indication more satisfaction with treatment.
Time Frame: End of treatment: approximately 3 months from intake
Population: Data is available for participants who attended post-treatment assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
score on a scale | 10.9 (1.3)

5. Secondary Outcome: Proportion of Participants Who Complete the Study Protocol
Description: Preliminary tolerability of the protocol will assessed by the number of enrolled participants who comply with all study procedures
Time Frame: End of treatment: approximately 3 months from intake
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 11
Participants | 10

6. Secondary Outcome: Change in Depressive Symptoms Over Time
Description: Change in symptoms as measured by the Hamilton Depression Rating Scale (HDRS-17; range 0-52) from pre- to post-treatment. Lower scores indicate better outcomes (reduction in symptoms).
Time Frame: At Baseline, At 4 weeks, Post-treatment: approximately 3 months from intake
Population: Treatment completers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
score on a scale
  Baseline | 17.27 (6.36)
  Midpoint (4 weeks) | 13.50 (4.50)
  Posttreatment | 10.10 (7.23)
Statistical Analysis 1: Comparison: Intervention; Test type: Other — ANOVA; p < 0.001, ANOVA; F ratio = 8.46 — The F ratio is used to evaluate the main effect of time in the ANOVA in relation to the critical F ratio. If it exceeds the critical F ratio, the null hypothesis (no effect of time) is rejected

7. Secondary Outcome: Change in Interoceptive Attention Style Over Time
Description: Changes in hypervigilance driven interoceptive attention and acceptance/mindfulness-based attention will be measured by the Multidimensional Assessment of Interoceptive Awareness (MAIA). The scale consists of 8 scales (addressing 5 dimensions of body awareness)The MAIA consists of 8 scales (addressing 5 dimensions of body awareness): Noticing (0-20); Not-Distracting (0-30); Not-Worrying (0-25); Attention Regulation (0-35); Emotional Awareness (0-25); Self-Regulation (0-20); Body Listening (0-15); Trust (0-15). A total scale score is not relevant. Higher scores indicate better outcomes (increased adaptive interoceptive attention).
Time Frame: Baseline, Post-treatment: approximately 3 months from intake
Population: Treatment completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
score on a scale
  Baseline: Noticing Subscale | 10.73 (3.13)
  Posttreatment: Noticing Subscale | 11.56 (3.57)
  Baseline: Not Distracting Subscale | 12.63 (5.30)
  Posttreatment: Not Distracting Subscale | 10.22 (4.29)
  Baseline: Not Worrying Subscale | 9.81 (2.18)
  Posttreatment: Not Worrying Subscale | 8.56 (2.79)
  Baseline: Attention Regulation Subscale | 15.73 (4.88)
  Posttreatment: Attention Regulation Subscale | 15.67 (4.15)
  Baseline: Emotional Awareness Subscale | 13.73 (3.64)
  Posttreatment: Emotional Awareness Subscale | 14.44 (4.07)
  Baseline: Self-Regulation Subscale | 7.00 (2.61)
  Posttreatment: Self-Regulation Subscale | 8.56 (2.65)
  Baseline: Body Listening Subscale | 5.00 (2.61)
  Posttreatment: Body Listening Subscale | 6.78 (2.17)
  Baseline: Trust Subscale | 5.18 (2.40)
  Posttreatment: Trust Subscale | 6.11 (2.76)

8. Secondary Outcome: Change in Cardiac Anxiety
Description: Change in cardiac anxiety from pre- to post-treatment assessment will be assessed using the Cardiac Anxiety Questionnaire (CAQ: score range: 0-72). Low scores mean better outcome (reduction in cardiac anxiety).
Time Frame: Baseline, Post-treatment: approximately 3 months from intake
Population: treatment completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
score on a scale
  Baseline | 36.67 (9.67)
  Posttreatment | 35.00 (10.39)

ADVERSE EVENTS:
Time Frame: Study duration (21 weeks)
Description: Our definition of adverse event and serious adverse event does not differ from the clinicaltrials.gov definition.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT04596891/Prot_SAP_000.pdf